CLINICAL TRIAL: NCT03498638
Title: Feasibility Study of Couple Therapy Treatment for Situational Couple Violence
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Keming Gao, Director, Mood Disorders Program, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9-13-27
Record Dates: First submitted 2018-03-30; First posted 2018-04-17 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Violence, Domestic
MeSH Terms: interventions — Couples Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couples Therapy (Experimental): Couples Therapy
  Interventions: Behavioral: Couples Therapy
- Control (Placebo Comparator): Couples Therapy after an 8 week waiting period
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Couples Therapy — Couples in the intervention group will receive couples therapy for 8 weekly sessions. Each therapy session will last approximately an hour. All therapies will be conducted by the PI, Dr. Gunnur Karakurt. Dr. Karakurt is a Licenced Marriage and Family Therapist and AAMFT (American Association of Marriage and Family Therapy) approved clinical supervisor. All therapies will be conducted as a couple. Training on stress management and safety planning will be performed as individuals. There will not be any group sessions. The goal of couple therapy is to help and improve couples' capacity to regulate emotions, solve problems, and communicate through therapy with the couple together.
  Arms: Couples Therapy
Other: Control — Couples in the control group will be taught safety planning, given information on local resources to help victims of violence, and will be instructed in stress and anger management strategies. Following this 8 week period, they will receive 8 weeks of couple therapy unless they choose not to.
  Arms: Control

SUMMARY:
The purpose of this study is to understand whether the couple therapy that is used in practice is effective in preventing situational couple violence. More specifically, investigators will focus on couples with mild to moderate forms of situational couple violence to investigate how couples therapy can be effective in preventing the escalation and recurrence of situational couple violence. For this purpose, the response of partners to therapy will be investigated by integrating self-report questionnaires and psycho-physiological markers of emotion.

ELIGIBILITY:
Inclusion Criteria:

* This study is open to married, dating, and cohabiting couples.
* Couples will have to be involved in an intimate relationship with their current partner for at least one year.
* Both partners have to be older than 18 years of age at the time they sign consent.
* Couples must have mild to moderate forms of situational couple violence.
* Both partners must want couples therapy and both partners must desire to maintain the relationship.
* Both individuals from the couple must participate concurrently, although they will sometimes be separated when asked questions of a sensitive nature.
* Only heterosexual couples will be included in the study.
* Both partners can be on psychotropic medication, if they are on medication and stable for past 12 month prior to enrollment, and no psychiatric hospitalization for past 2 years.

Exclusion Criteria:

* Couples will be excluded from the study if there are indicators of severe intimate partner violence and/or characterological violence as this study targets couples with mild to moderate levels of violence. In order to distinguish between these two different types of violence, we will use specific items in the Conflict Tactic Scale (CTS) completed by both parties (Johnson, & Leone, 2005). Severe and/or characterological violence in this study is defined as follows:

  * If participants answer yes to both of the following items: "I punched or hit my partner with something that could hurt", "I kicked my partner".
  * If participants answer yes to any of the following items: "I choked my partner," "I slammed my partner against a wall," "I beat up my partner" "I burned or scalded my partner on purpose," and "I used a knife or gun on my partner".
  * One of the partners reports that a violent behavior was repeated at least six times in a year by their partner or themselves.
* Participants will also be excluded from the study if they answer yes to the following questions: "Do you have any firearms at home?", "In your previous relationships, did your partners ever tell you that you were physically abusive?"
* Participants will be excluded from the study if they are not stable on psychiatric medication for more than 12 months.
* Couples will be excluded from the study if there is a discrepancy between partners' reports of violence (received or perpetrated) in the CTS, defined as the difference between the partners' reports of the frequency of a particular act by the same partner. If the difference of the average score of the partners, or for any of the acts in the scale in the CTS is greater than 2, the couple will be excluded from the study. For example, if the female partner reports that the male partner pushed her three times but the male partner reports that he never pushed his partner, the couple will be excluded from the study since the couple will receive a difference score of three for the act of pushing.
* Participants will be excluded from the study if undiagnosed, untreated serious mental illness is suspected during pre-screening. In order to screen participants with severe mental health problems, Symptom Checklist (SCL90) will be used. We will use the cut off 0.885 with the area under the receiver operating characteristic (ROC) curve with lower and upper bounds of the 95% confidence interval.
* Participants will be excluded from the study if there are indicators of substance misuse. We will use the 16 item Simple Screening Instrument for Substance Abuse (SSISA) to screen participants' substance use. We'll score only 14 items out of the 16 items, which were selected by the Treatment Improvement Protocols (TIP) 11 consensus panelists from existing alcohol and drug abuse screening tools. A score of 4 or greater has become the established cutoff point.
* Participants will be excluded if they reported any history of violent legal offences in the past 2 years.
* Participants will be excluded if participants are currently suicidal and/or psychotic and/or patients who is moderately ill (e.g. equivalent of Clinical Global Impression (CGI) score 3 or greater) at the pre-screening.
* Participants who are not literate or cannot speak English will be excluded. The questionnaires require a 6th grade reading level.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01-19 (Actual); Primary Completion 2017-05-24 (Actual); Study Completion 2017-05-24 (Actual)

PRIMARY OUTCOMES:
Association between change in Intimate Partner Violence (IPV) and change each partner's psychophysiological regulation in terms of Hypothalamic Pituitary Adrenal (HPA) activity | Baseline and Week 8
  This aim will investigate whether dysregulation of HPA activity in each partner is correlated with the existence and intensity of IPV for the couple. HPA activity will be measured using salivary cortisol.
Examine the associations between change IPV and change each partner's psychophysiological regulation in terms of Parasympathetic Nervous System (PNS) activity. | Baseline and Week 8
  This aim will investigate whether dysregulation of PNS activity in each partner is correlated with the existence and intensity of IPV for the couple. PNS activity will be measured using vagal tone and vagal regulation by using an eMotion Heart Rate Variability (HRV) sensor.

SECONDARY OUTCOMES:
Examine the longitudinal effects of conjoint therapy on IPV and each partner's psychophysiological regulation in terms of HPA | Baseline and Week 8
  In couples where IPV decreases, this aim will investigate whether that decrease in IPV is correlated with a change in regulation of HPA activity for each partner.
Examine the longitudinal effects of conjoint therapy on IPV and each partner's psychophysiological regulation in terms of PNS activity | Baseline and Week 8
  In couples where IPV decreases, this aim will investigate whether that decrease in IPV is correlated with a change in regulation of PNS activity for each partner.
Examine the correlation between one partner's psychophysiological regulation as measured by HPA activity between the other partner's HPA activity. | Baseline and Week 8
Examine the correlation between one partner's psychophysiological regulation as measured by PNS activity between the other partner's PNS activity. | Baseline and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Gunnur Karakurt, PhD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03498638/Prot_SAP_000.pdf